CLINICAL TRIAL: NCT04146246
Title: Comparative Evaluation of the FINDERTM Instrument and FINDERTM G6PD Cartridge in Adults and Neonates
Brief Title: Comparative Evaluation of the FINDER Instrument and FINDER G6PD Cartridge in Adults and Neonates
Status: Completed | Type: Observational
Sponsor: Baebies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSPROJ00004001
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: G6PD; G6PD Deficiency
Keywords: G6PD; Neonate
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Adult: Adults aged 18 years or older. Collect whole blood sample via venous/arterial puncture and, where possible, finger stick.
  Interventions: Diagnostic Test: G6PD assay
- Neonate: Neonates gestational age >35 weeks or older. Collect whole blood sample via heel prick or, where an in dwelling line already exists, via arterial/umbilical draw.
  Interventions: Diagnostic Test: G6PD assay

INTERVENTIONS:
Diagnostic Test: G6PD assay — A test for G6PD deficiency.

SUMMARY:
A prospective clinical study to compare the clinical performance of the FINDER™ Instrument and the G6PD assay to an FDA cleared instrument/reagent combination in adult and neonate populations.

DETAILED DESCRIPTION:
A prospective clinical study to compare the clinical performance of the FINDER™ Instrument and the G6PD assay to an FDA cleared instrument/reagent combination in adult and neonate populations. Neonate and adult subjects will be recruited from 3 clinical sites. Neonate samples will be collected as heel prick unless an in dwelling line is already in place at which point a venous or arterial/umbilical sample will be collected. Adult samples will be collected as venous/arterial samples and finger stick samples. Samples will be tested at the point of care/near patient and in the clinical laboratory using the FINDER Instrument and G6PD assay on a digital microfluidic platform. Samples will also be sent to a third party CLIA laboratory for test using an FDA 510(k) cleared instrument/reagent combination for G6PD.

ELIGIBILITY:
Inclusion Criteria:

* Neonates aged >35 gestational weeks or older.
* Adult subjects who are age 18 and older.
* Adult subjects who weigh at least 110 pounds.
* All ethnicities.
* Male and female subjects.

Exclusion Criteria:

* Adult subjects who weigh less than 110 pounds.
* Subjects with anemia for which an attending physician will not authorize a blood draw.
* Subjects who have received a blood transfusion.
* Subjects who are pregnant.

Ages: 35 Weeks to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults who are at least 18 years of age or older. Neonates who are at least 35 gestational weeks old, recruited from the well baby nursery or the NICU.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
G6PD enzymatic activity in adults and neonates | Immediately following a blood draw.
  G6PD enzymatic activity in the FINDER System for adults and neonates compared to the G6PD activity tested using a known FDA cleared assay/instrument combination

SECONDARY OUTCOMES:
Point of care/near patient results and clinical laboratory results | Immediately following a blood draw.
  Characterization of the performance of the FINDER device when used at a POC/near patient location and when used in a clinical laboratory location.
Arterial/venous whole blood results and tissue capillary test results | Immediately following a blood draw.
  Characterization of the performance of the FINDER G6PD assay when tested with blood from a venipuncture or arterial puncture, including umbilical catheter access, and where possible, performance will be evaluated when tested with blood from tissue puncture capillary samples.

CONTACTS AND LOCATIONS:
Overall Officials: Rama Sista, PhD, Study Director — Director Product Development
Locations (3):
- United States (3):
  - Duke Health, Durham, North Carolina
  - Wake Med, Raleigh, North Carolina
  - University Hospitals Cleveland Medical Center Rainbow Children's Hospital, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No